CLINICAL TRIAL: NCT07393581
Title: Group Music Therapy, Emotional Well-Being, Health, and Social Connectedness Among University Students in Urban China: A Randomized Controlled Trial
Brief Title: Group Music Therapy for Emotional Well-Being and Social Connectedness
Acronym: GMT2025
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Yangzhou University (Other)
Responsible Party: Principal Investigator, Ling Yang, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GMT2025
Record Dates: First submitted 2026-01-28; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Emotional Well-Being; Social Connectedness
Keywords: group music therapy; active music therapy; receptive music therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Music Therapy (MT-A) (Experimental): Weekly in-person active group music therapy sessions for 6 weeks (60 minutes per session; groups of 10-15 participants) facilitated by trained music therapists. Sessions included group singing, rhythmic improvisation using body percussion or simple instruments, collaborative musical games, and brief guided group discussion.
  Interventions: Behavioral: Active Group Music Therapy
- Receptive Music Therapy (MT-R) (Experimental): Weekly in-person receptive group music therapy sessions for 6 weeks (60 minutes per session; groups of 10-15 participants) facilitated by trained music therapists. Sessions included guided music listening, music-assisted imagery/visualization, reflective writing or moderated discussion, and breathing/relaxation exercises.
  Interventions: Behavioral: Receptive Group Music Therapy
- Waitlist Control (No Intervention): Participants received no sessions during the 6-week study period and completed baseline and post-intervention assessments. After study completion, participants were offered the option to attend one group music therapy session.

INTERVENTIONS:
Behavioral: Active Group Music Therapy — Active group music therapy delivered in person once weekly for 6 weeks (60 minutes per session). Activities included group singing, rhythmic call-and-response, body percussion, simple percussion instruments, and collaborative musical games.
  Arms: Active Music Therapy (MT-A)
Behavioral: Receptive Group Music Therapy — Receptive group music therapy delivered in person once weekly for 6 weeks (60 minutes per session). Activities included guided music listening, music-assisted imagery/visualization, reflective writing or moderated discussion, and breathing/relaxation exercises.
  Arms: Receptive Music Therapy (MT-R)

SUMMARY:
This randomized controlled trial evaluated whether two formats of group music therapy can improve emotional well-being, self-rated health, and social connectedness among undergraduate students living in urban areas in China. A total of 120 students were randomly assigned to one of three conditions: (1) active group music therapy, (2) receptive group music therapy, or (3) a waitlist control group.

Both music therapy programs were delivered in person over 6 weeks, with one 60-minute session per week facilitated by trained music therapists. The active format emphasized participatory music-making (e.g., singing, rhythmic activities, and group improvisation), while the receptive format focused on guided music listening and reflection.

Participants completed self-report questionnaires at baseline and immediately after the 6-week period assessing positive and negative affect, anxiety symptoms, general health, and perceived social connectedness. The study examined whether the two music therapy approaches led to improvements compared with the waitlist control condition.

DETAILED DESCRIPTION:
This study used a parallel-group randomized controlled design to examine the effects of two structured formats of group music therapy on emotional well-being, anxiety symptoms, self-rated health, and social connectedness among undergraduate students in urban China. Participants were recruited through university announcements and campus-based advertisements. Eligible participants provided informed consent and completed baseline assessments before being randomly allocated to one of three conditions: active group music therapy, receptive group music therapy, or a waitlist control group.

The intervention period lasted 6 weeks. Participants assigned to either music therapy condition attended weekly in-person group sessions of approximately 60 minutes in small groups (10-15 participants). Sessions were delivered by trained music therapists using standardized protocols to ensure structural equivalence across conditions. The active group music therapy format emphasized participatory music-making (e.g., group singing, rhythmic call-and-response, body percussion, and collaborative musical activities) and included brief guided group discussion at the end of each session. The receptive group music therapy format emphasized guided music listening, music-assisted imagery/visualization, reflective writing or moderated discussion, and relaxation/breathing exercises.

Participants in the waitlist control condition did not receive any intervention during the 6-week study period but completed the same baseline and post-intervention assessments as the intervention groups. After completion of the study, waitlist participants were offered the option to attend one group music therapy session.

All outcomes were assessed using self-report measures administered at baseline and immediately after the 6-week period.

ELIGIBILITY:
Inclusion Criteria:

Undergraduate university students aged 18 to 26 years

Living in an urban area in China

Able to attend weekly in-person group sessions for 6 weeks

Provided written informed consent

Exclusion Criteria:

Self-reported severe active clinical diagnosis

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms (GAD-7 total score) | Baseline (pre-intervention) and immediately post-intervention (6 weeks)
  Anxiety symptoms assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7). Higher scores indicate greater anxiety severity.

SECONDARY OUTCOMES:
Positive affect (I-PANAS-SF Positive Affect subscale) | Baseline (pre-intervention) and immediately post-intervention (6 weeks)
  Positive affect assessed using the International Positive and Negative Affect Schedule Short Form (I-PANAS-SF), Positive Affect subscale. Higher scores indicate higher positive affect.
Negative affect (I-PANAS-SF Negative Affect subscale) | Baseline (pre-intervention) and immediately post-intervention (6 weeks)
  Negative affect assessed using the International Positive and Negative Affect Schedule Short Form (I-PANAS-SF), Negative Affect subscale. Higher scores indicate higher negative affect.
Self-rated general health (SF-36 General Health subscale) | Baseline (pre-intervention) and immediately post-intervention (6 weeks)
  General health assessed using the Short Form Health Survey (SF-36), General Health subscale. Scores are transformed to a 0-100 scale, with higher scores indicating better perceived health.
Social connectedness (Social Connectedness Scale-Revised) | Baseline (pre-intervention) and immediately post-intervention (6 weeks)
  Social connectedness assessed using the Social Connectedness Scale-Revised (SCS-R), Social Connectedness subscale. Higher scores indicate stronger perceived social connectedness.

CONTACTS AND LOCATIONS:
Locations (1):
- Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data and study materials will be made publicly available via the Open Science Framework (OSF).
Supporting Information: Study Protocol, Analytic Code
Time Frame: De-identified IPD and supporting information will be available immediately following publication and will remain available indefinitely.
Access Criteria: De-identified individual participant data and supporting information will be publicly available to anyone via the Open Science Framework (OSF). No application or data use agreement will be required.
URL: https://osf.io/nkmt8/?view_only=3ac94bba48664cb1aaedf0d1f799377c

REFERENCES:
- See also: Open Science Framework (OSF) page with study materials and de-identified data for this trial. — https://osf.io/nkmt8/?view_only=3ac94bba48664cb1aaedf0d1f799377c
- Available data/document: Individual Participant Data Set: OSF — https://osf.io/nkmt8/?view_only=3ac94bba48664cb1aaedf0d1f799377c — De-identified participant-level data and supporting information are available via the Open Science Framework (OSF).
- Available data/document: Study Protocol: OSF — https://osf.io/nkmt8/?view_only=3ac94bba48664cb1aaedf0d1f799377c — Study protocol and intervention materials available on OSF.